CLINICAL TRIAL: NCT06160349
Title: EnCoRe MoMS Aim 3: Engaging Communities to Reduce Morbidity From Maternal Sepsis
Brief Title: EnCoRe MoMS: Engaging Communities to Reduce Morbidity From Maternal Sepsis (Aim 3)
Status: Enrolling by invitation | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Northern Manhattan Perinatal Partnership (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dena Goffman, Ellen Jacobson Levine and Eugene Jacobson Professor of Women's Health (in Obstetrics and Gynecology), Columbia University
Other Study IDs: AAAU3697 - Aim 3; 1UG3HD111247 (NIH)
Record Dates: First submitted 2023-11-20; First posted 2023-12-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Maternal Sepsis; Infections
Keywords: Post Partum Period; Pregnancy; Maternal Health; Electronic Health Record
MeSH Terms: conditions — Pregnancy Complications, Infectious; Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Interviews: Patients with risk factors for maternal sepsis interviewed about pregnancy, labor/delivery, and postpartum via Zoom.
- Community Stakeholders: Community stakeholders with professional and/or academic backgrounds relevant to maternal health who participate in focus group discussion.

SUMMARY:
Sepsis is the second leading cause of maternal death in the U.S. For racial and ethnic minoritized birthing people, especially those who are Black, living in poverty, and from underserved communities, labor and postpartum are particularly vulnerable risk periods. The goal of this multi-center, multidisciplinary observational study is to establish a novel maternal care continuity model to reduce sepsis- related death and disability and increase maternal health equity.

DETAILED DESCRIPTION:
Maternal sepsis is the second leading cause of maternal death, major cause of morbidity, and preventable in most cases. Labor, birth, and postpartum are periods of increased sepsis risk, particularly for racial and ethnic minoritized birthing people. With extensive community partnerships and community organized leadership advisory board (CoLAB), EnCoRe MoMS: Engaging Communities to Reduce Morbidity from Maternal Sepsis (Aim 3) Conduct a co-design process and qualitative study to explore the experiences, needs, and perceived solutions for maternal care continuity, sepsis prevention, and promotion of equity in postpartum.

In the UG3 phase, robust community engagement and research infrastructures were established to: 3a. (3a.1) Refine the CoLAB and co-design process; (3a.2) Conduct in-depth individual patient interviews (IDIs) and focus group discussions (FGDs) with community and hospital stakeholders from one site to explore the lived experiences and perspectives of SDOH on care access/quality, outcome disparities, and solutions for care continuity.

In the UH3 phase, the investigators will engage the community toAim 3b. (3b.1) Complete qualitative patient IDIs and stakeholder FGDs for the three additional hospital sites; (3b.2) Co-design an integrative supportive care model, with our community partner co-lead, CoLAB, and results from other aims, that entails maternal sepsis community engagement, care linkages, education, services, and policy efforts. The resulting model can be scaled to hospitals and communities with lesser resources and applied to other preventable causes of severe maternal morbidity.

ELIGIBILITY:
Inclusion Criteria:

Patient Interviews:

* Speak Spanish or English
* Be 18 years or older
* Have a birthing experience in Columbia, Allen, Lincoln, or Harlem Hospitals within the past 8 weeks of enrollment
* Have had at least one early warning sign or risk factor for infection present during their pregnancy, delivery, or postpartum

Community Stakeholder Focus Groups:

* Speak English or Spanish
* Be 18 years or older
* Have academic/professional background relevant to maternal health in New York City.

Exclusion Criteria:

Patient Interviews

* Under 18 years old
* Speaks a language other than Spanish or English
* Gave birth in a hospital other than Columbia, Allen, Lincoln, or Harlem Hospitals
* Did not have had at least one early warning sign or risk factor for infection present during their pregnancy, delivery, or postpartum

Community Stakeholder Focus Groups

* Under 18 years old
* Speaks a language other than Spanish or English
* Does not have a academic/professional background relevant to maternal health in New York City.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For patient interviews- Adult women have a birthing experience in Columbia, Allen, Lincoln, or Harlem Hospitals within the past 8 weeks of enrollment
  For focus groups- stakeholders with academic/professional backgrounds relevant to maternal health
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Integrative Supportive Care Model | 2023-2025
  Patient and community stakeholder feedback regarding lived experiences and perspectives of the impact of SDOH on care access and quality will be assessed by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Dena Goffman, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Columbia Unviersity Medical Center, New York, New York
  - NYC Health+Hospitals/Harlem, New York, New York
  - NYC Health + Hospitals/Lincoln, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No